CLINICAL TRIAL: NCT03484676
Title: Adequacy of One-Point Fixation of Displaced Zygomatic Complex Fractures Using a Customized Plate pre_post Study
Brief Title: Adequacy of One Point Fixation of Displaced Zygomatic Complex Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Ashour Saad Borma, Internal resident at Maxillofacial department, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-03-17
Record Dates: First submitted 2018-03-13; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Zygomatic Fractures
MeSH Terms: conditions — Zygomatic Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unilateral Non comminuted zygomatic complex fracture (Other): Patient undergo treatment no control group
  Interventions: Device: Titinium

INTERVENTIONS:
Device: Titinium — custom made plate at one point after 3D virtual simulation and reduction of the complex using Mimics software.

SUMMARY:
Patients with unilateral non-comminuted zygomatic complex fracture undergo fixation of the complex by a customized plate at one point after 3D virtual simulation and reduction of the complex using Mimics software.

DETAILED DESCRIPTION:
History data will be gathered including personal data, medical and surgical history, and family history.

Clinical examination and photographic records will be carried out to evaluate the magnitude and direction of the displaced zygoma, degree of facial asymmetry, neurosensory affection and functional disturbances.

Computed tomography (CT) scan:

Patients will receive a preoperative computed tomography (CT) scan of the facial bones [ Axial cuts, DICOM file, Gantry tilt zero and minimal thickness of 1 mm]. The radiographic data will be imported into a surgical simulation software to virtually reduce the fractured zygoma and custom design the plate for fixation.

General operative procedures:

* All cases will undergo surgery under general anesthesia with nasotracheal intubation.
* Intraoral maxillary vestibular approach will be used to gain access to the fractured zygomatic complex. Reduction of the fractured segment would be achieved using the appropriate techniques and instrumentation. One point ORIF would be accomplished using the customized plate.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age range from 15-65 years.
* Patients with unilateral zygomatic complex fracture
* Displaced fracture
* Dentulous or edentulous patients.
* Patients should be free from any systemic disease that may affect normal healing of bone and predictable outcome.

Exclusion Criteria. Patients with systemic diseases as history of radiation therapy or chemotherapy, hematological disorders, neuromotor disorders and autoimmune diseases (may affect normal healing).

* Patients with comminuted fractures .
* Delayed presentation 3 weeks or more after the date of trauma.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction. Measuring device visual analogue scale. Measuring unit 0-10 | One week
  Esthetics and function of patient return post operative. Normal

SECONDARY OUTCOMES:
Adequacy of reduction compared to the preoperative virtual simulation measuring device mimics software Ware. Measuring unit millimeters | Immediately post operative
  Reduction of fracture on mimics soft ware depending on 3d virtual simulation and mirror image of the same patient and after operation I will compare post operative reduction to preoperative reduction on mimics soft ware in millimeters measuring unit